CLINICAL TRIAL: NCT03629587
Title: Helicobacter Pylori and it's Hematological Impact
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Mohamed Mahmoud, Demonstrator at internal medicine department, principle investigator, Assiut University
Other Study IDs: H pylori
Record Dates: First submitted 2018-07-15; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: H Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histopathological tissues and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients presented H pylori positive: Upper endoscopy, Gastric biopsy, CBC, VITAMIN B12 level, iron studys, folic acid level, bone marrow aspirate
- Patients with H pylori negative: Upper endoscopy, Gastric biopsy, CBC, VITAMIN B12 level, iron studys, folic acid level, bone marrow aspirate

SUMMARY:
To evaluate the effect of helicobacter pylori on the blood for proper management

DETAILED DESCRIPTION:
r pylori (H. pylori)is the most common infection in humans, with a marked disparity between developed and developing countries.It presents in over 50% of all stomachs in the world population, making it the most frequent infection in humanS. It displays a marked disparity in occurrence between developed countries, where its prevalence oscillates between 30% and 50%, and developing countries, where its prevalence ranges between 80% and 90%.

Although H. pylori infections are asymptomatic in most infected individuals, they are intimately related to malignant gastric conditions such as gastric cancer and gastric mucosa-associated lymphoid tissue (MALT) lymphoma and to benign diseases such as gastritis and duodenal and gastric peptic ulcers.

Since it was learned that bacteria could colonize the gastric mucosa, there have been reports in the medical literature of over 50 extragastric manifestations involving a variety medical areas of specialization. These areas include cardiology, dermatology, endocrinology, gynecology and obstetrics, hematology, pneumology, odontology, ophthalmology, otorhinolaryngology and pediatrics, and they encompass conditions with a range of clear evidence between the H. pylori infection and development of the disease.

This review focuses on hematologic diseases included in international consensus and management guides for H. pylori infection; specifically iron deficiency Anemia, vitamin B12 (cobalamin) deficiency, immune thrombocytopenia, and extranodal marginal zone mucosa-associated lymphoid tissue lymphoma (MALT Lymphoma). In addition of other hematologic diseases not included in guides and consensus as auto-immune neutropenia, antiphospholipid syndrome, and plasma cell dyscrasias.

Iron deficiency Iron deficiency (ID) is a serious public health issue, regardless of whether it is associated with anemia . It is especially important to remember that ID is a chronic process with a slow onset, in which the iron imbalance may take several years to establish and manifest clinically. One of the consequences can be observed through blood characteristics such as morphological alterations of erythrocytes or the presence of anemia, according to the criteria of the WHO.ID occurs in three stages: pre-latent (stage 1), in which ferritin is between 12 and 30 μg/L, latent (stage 2) when the ferritin falls below 12 μg/L, and ID anemia (stage 3) when anemia is present in addition to diminished or depleted reservoir iron levels (determined by serum ferritin).

Vitamin B12 deficiency Vitamin B12 is required as a coenzyme for the metabolism of the amino acids methionine, threonine and valine and for the transformation of methyl-tetrahydrofolate to tetrahydrofolate, which is necessary for DNA synthesis. Vitamin B12 deficiency, also known as cobalamin deficiency, is defined by low serum values of vitamin B12 and both homocysteine and methylmalonic acid (two components of the vitamin B12 metabolic pathway). Vitamin B12 deficiency occurs as a result of antibodies directed against gastric parietal cells and intrinsic factor, in addition to achlorhydria and a decrease in pepsinogen I and gastrin.

The laboratory diagnosis of vitamin B12 deficiency is established in accordance with the following criteria:

1. serum vitamin B12 levels < 150 pmol/L (< 200 pg/mL) with clinical features and/or hematological anomalies related to vitamin B12 deficiency
2. serum vitamin B12 levels < 150 pmol/L on two separate occasions .
3. serum vitamin B12 levels < 150 pmol/L and total serum homocysteine levels > 13 μmol/L or methylmalonic acid levels > 0.4 μmol/L (in the absence of renal failure and folate and vitamin B6 deficiencies).
4. serum holotranscobalamin levels < 35 pmol/L. Immune thrombocytopenia Primary immune thrombocytopenia (ITP), previously called idiopathic thrombocytopenic purpura and autoimmune thrombocytopenic purpura.ITP has been redefined as "an autoimmune disorder characterized by isolated thrombocytopenia (peripheral blood platelet count 100 × 109/L) in the absence of other causes or disorders that may be associated with thrombocytopenia.

Primary ITP is associated with congenital or acquired immune disorders, leading to an autoimmune response against platelets or megakaryocytes and characterized because it is not associated with other alterations.

Gastric MALT lymphoma Gastric MALT lymphoma is a rare form of non-Hodgkin lymphoma that affects B lymphocytes and typically develops in lymphoid tissue associated with mucous membranes and rarely in lymph nodes. It represents approximately 5% of all diagnosed non-Hodgkin lymphomas.

The mechanisms by which H. pylori produces the appearance of a lymphoma similar to gastric carcinogenesis has not been fully clarified, but it is likely that environmental, host, and bacterial-related factors must be involved.H. pylori infection leads to development of MALT lymphoma and can take the following course. First, the infection gives rise to a lymphocyte response that conditions a polyclonal B lymphocyte response and MALT formation through antibody production. Then, different lymphocyte populations would maintain the response provoked by the bacteria. In the polyclonal MALT proliferation, a monoclonal population of B-cells could appear and accumulate cytogenetic changes such as translocations, mutations, microsatellite instabilities, eventually evolving into a low-grade MALT lymphoma that is dependent on H. pylori-related antigen stimuli. Finally, new cytogenetic changes such as translocations, suppressor gene deactivation (p53 and p16, among others), and c-myc activation would make this neoplastic population of monoclonal B-cells escape from its dependence on T lymphocytes and H. pylori antigens and favor its transformation into a high-grade lymphoma. As a result of this sequence of events, a low- or high-grade lymphoma would ultimately develop.

UNRECOGNIZED HEMATOLOGIC MANIFESTATIONS This group includes autoimmune neutropenia, antiphospholipid syndrome, plasma cell dyscrasia including monoclonal gammopathy of undetermined significance and multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* All patients complained of symptoms suggestive of gastritis whether acute (within two weeks) or chronic (three or more months) and were diagnosed at endoscopy to have H.pylori infection by biopsy.
* Patients aged more than 18 years old.
* Both sexes (male & female).

Exclusion Criteria:

* Patients with malignant diseases or Gastric malignancy.
* Other causes of Thrombocytopenia as systemic lupus erythematous and human immunodeficiency virus and or acquired immunodeficiency syndrome.
* Other causes of Anemias with or without blood loss.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 patients were presented with symptoms suggesting of gastritis, Group (A) 50 patients with positive H .Pylori biopsy, Group (B): 50 patients with negative H.pylori biopsy.
  All patients and control group were submitted to:1- Detailed history of age, sex, associate diseases, and family history of the same illness or others.2- Detailed history about gastric symptoms and duration of the disease 3-Full clinical examination 4- Laboratory investigations including:
  * Complete blood count with reticulocytic count.- Upper endoscopy - Diagnostic biopsy
  * Serum iron, total iron binding capacity and serum Ferritin.- Vitamin B 12 and folic acid level if indicated- Bone marrow aspirate if indicated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Upper endoscopy | 2 year
  To demonstrate infection of H PyloruPylorifohistopathological examination

SECONDARY OUTCOMES:
Complete blood count | 2 year
  to assess type of anemia and hematological affection
Iron studies | 2 year
  To assess iron deficiency anemia
Vitamin B 12 level and folic acid level | 2 year
  To demonstrate level of vitamin B12
Bone marrow aspiration | 2 year
  To determine other causes of bone marrow affection

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fischbach W, Malfertheiner P. Helicobacter Pylori Infection. Dtsch Arztebl Int. 2018 Jun 22;115(25):429-436. doi: 10.3238/arztebl.2018.0429. PMID 29999489
- [Background] Martinson HA, Shelby NJ, Alberts SR, Olnes MJ. Gastric cancer in Alaska Native people: A cancer health disparity. World J Gastroenterol. 2018 Jul 7;24(25):2722-2732. doi: 10.3748/wjg.v24.i25.2722. PMID 29991877
- [Background] Fukuda T, Asou E, Nogi K, Yasuda M, Goto K. Association between Helicobacter pylori infection and platelet count in mice. Exp Anim. 2018 Nov 1;67(4):487-492. doi: 10.1538/expanim.18-0004. Epub 2018 Jun 7. PMID 29877197
- [Background] Best LM, Takwoingi Y, Siddique S, Selladurai A, Gandhi A, Low B, Yaghoobi M, Gurusamy KS. Non-invasive diagnostic tests for Helicobacter pylori infection. Cochrane Database Syst Rev. 2018 Mar 15;3(3):CD012080. doi: 10.1002/14651858.CD012080.pub2. PMID 29543326
- [Background] Barbosa AMC, Ribeiro RA, Silva CISM, Cruz FWS, Azevedo OGR, Pitombeira MHDS, Braga LLC. Platelet count response to Helicobacter pylori eradication for idiopathic thrombocytopenic purpura in northeastern Brazil. Hematol Transfus Cell Ther. 2018 Jan-Mar;40(1):12-17. doi: 10.1016/j.bjhh.2017.09.005. Epub 2017 Nov 24. PMID 29519366
- [Background] Kim H, Lee WS, Lee KH, Bae SH, Kim MK, Joo YD, Zang DY, Jo JC, Lee SM, Lee JH, Lee JH, Kim DY, Ryoo HM, Hyun MS, Kim HJ; CoOperative Study Group A for Hematology (COSAH). Efficacy of Helicobacter pylori eradication for the 1st line treatment of immune thrombocytopenia patients with moderate thrombocytopenia. Ann Hematol. 2015 May;94(5):739-46. doi: 10.1007/s00277-014-2268-9. Epub 2014 Dec 13. PMID 25501820
- [Background] Papagiannakis P, Michalopoulos C, Papalexi F, Dalampoura D, Diamantidis MD. The role of Helicobacter pylori infection in hematological disorders. Eur J Intern Med. 2013 Dec;24(8):685-90. doi: 10.1016/j.ejim.2013.02.011. Epub 2013 Mar 21. PMID 23523153
- [Background] Jafarzadeh A, Akbarpoor V, Nabizadeh M, Nemati M, Rezayati MT. Total leukocyte counts and neutrophil-lymphocyte count ratios among Helicobacter pylori-infected patients with peptic ulcers: independent of bacterial CagA status. Southeast Asian J Trop Med Public Health. 2013 Jan;44(1):82-8. PMID 23682441